CLINICAL TRIAL: NCT06413979
Title: Testing the Feasibility of a Family-based Adjunctive Treatment Protocol for Targeting Co-Occurring Internalizing Disorders Among Adolescents with SUD
Brief Title: Family Support Protocol for Adolescent Internalizing Disorders
Acronym: Fam-AID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA056026 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Internalizing Disorders; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Interrupted Time Series Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fam-Aid (Experimental)
  Interventions: Behavioral: Family Support Protocol for Adolescent Internalizing Disorders (Fam-AID)

INTERVENTIONS:
Behavioral: Family Support Protocol for Adolescent Internalizing Disorders (Fam-AID) — (1) Family Engagement of caregivers and primary supports in treatment planning and services; (2) Relational Reframing of family constraints, resiliencies, and social capital connected to the youth's ID symptoms; (3) Functional Analysis of the youth's ID symptoms and related behaviors; (4) Cognitive-behavioral therapy (CBT) core techniques to address the youth's ID symptoms and functional needs, featuring three transdiagnostic interventions (emotion acceptance, emotional exposure, behavioral activation) to address negative affect and emotional dysregulation underlying both depression and anxiety; and (5) Family Psychoeducation and Safety Planning focused on education about comorbid SUD/ID and prevention of youth self-harm. All interventions featured in each module have strong empirical support.

SUMMARY:
This R34 will develop and test an adjunctive treatment protocol for addressing co-occurring internalizing disorders among adolescents enrolled in usual care for substance use problems. Internalizing disorders (ID), primarily depression and anxiety, are highly prevalent among youth receiving community-based treatment for substance use disorder (SUD). Comorbidity rates range from 30-70% due to the multiple developmental pathways by which adolescent SUD and ID cause and exacerbate one another. Moreover, unresolved ID issues significantly interfere with youth SUD treatment and recovery processes. Yet, the youth SUD clinical workforce is not systematically educated or trained in evidence-based practices for ID; thus, line services for youth SUD do not systematically target ID. The research literature offers a few integrated behavioral models for simultaneously treating both SUD and ID in youth; however, such models feature intensive manualized procedures that have proven cumbersome to scale and deliver in frontline settings. As a result, the clinical workforce, though desiring ID-focused training, currently has inadequate resources for treating ID effectively.

A promising solution to diminish this quality gap is developing an adjunctive, modular protocol to augment routine care for comorbid SUD/ID by directly targeting ID as a key treatment goal: Family Support Protocol for Adolescent Internalizing Disorders (Fam-AID). As an adjunctive protocol, Fam-AID will not require clinicians to markedly alter existing base practices for SUD. It will be anchored by three evidence-based foundations for treating co-occurring adolescent ID. First, it prioritizes family engagement in services and family-oriented treatment goals, which have been shown to enhance outcomes for youth SUD and ID alike. Second, it is a modular protocol that features core elements of manualized treatment for ID; core element interventions enhance treatment effectiveness by fostering implementation feasibility and sustainability in usual care. Third, it seeks to reinforce the family safety net to prevent teen self-harm. In accord with these foundations, and pending pilot development, we anticipate that Fam-AID will contain five treatment modules that can be delivered in any sequence to meet client needs: (1) Family Engagement of caregivers and primary supports in treatment planning and services; (2) Relational Reframing of family constraints, resiliencies, and social capital connected to the youth's ID symptoms; (3) Functional Analysis of the youth's ID symptoms and related behaviors; (4) Cognitive-behavioral therapy (CBT) core techniques to address the youth's ID symptoms and functional needs, featuring three transdiagnostic interventions (emotion acceptance, emotional exposure, behavioral activation) to address negative affect and emotional dysregulation underlying both depression and anxiety; and (5) Family Psychoeducation and Safety Planning focused on education about comorbid SUD/ID and prevention of youth self-harm. All interventions featured in each module have strong empirical support.

The Fam-AID protocol will contain several innovations intended to boost treatment feasibility and impact for this vulnerable group. Aligned with the core elements strategy, it will be designed for uptake by all motivated clinicians regardless of their clinical orientation and training. It will use evidence-based family engagement techniques to systematically integrate caregivers in the treatment process; typically, families are not centralized in SUD services for youth despite compelling empirical and clinical rationale to do so. It will feature a treatment customization exercise in which clients and therapists collaboratively select CBT techniques to integrate in ongoing treatment based on functional ID assessment.

To achieve study aims we will first develop a Fam-AID implementation toolkit during a three-part Pilot Phase at one pilot site: (a) Solicit provider input on Fam-AID components; (b) Create video-based training and fidelity procedures, leveraging the PI's existing online therapist training and consultation resources in core CBT techniques for adolescent SUD, as well as the Co-I's equivalent training resources for adolescent ID; (c) Pilot the toolkit with 4-6 clients. In Years 2-3 we will conduct an Interrupted Time Series Study for N = 60 SUD/ID cases across two sites serving diverse youth: 30 will receive TAU, and then following line staff training, 30 new cases will receive TAU enhanced by adjunctive Fam-AID. Aim 1: Feasibility will examine Fam-AID cases for acceptability via client and therapist interviews and fidelity benchmarks via therapist- and observer-report of module coverage and protocol dose. Aim 2: Outcomes will test TAU vs. TAU + Fam-AID for immediate impact on family member attendance and ultimate impacts on adolescent ID symptoms at 3- and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Youth is age 13-21.
* Youth lives with a primary caregiver who can attend treatment sessions.
* Youth endorses one or more DSM-5-TR symptoms for SUD and meets American Society of Addiction Medicine criteria for outpatient SU treatment.
* Youth meets DSM-5-TR criteria, or has elevated symptoms and impairment, for any of the following IDs: Current or Recurrent Major Depressive Episode, Pervasive Depressive Disorder, Social Anxiety Disorder, Generalized Anxiety Disorder, Panic Disorder, Posttraumatic Stress Disorder.
* Youth completes intake and is enrolled as an active case at study site

Exclusion Criteria:

* Illness requiring hospitalization
* Current psychotic symptoms
* Severe SU problems that require immediate relief (detox or residential placement)
* Pervasive developmental disorder.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Fidelity | Baseline to 6 months follow-up
  Therapist and observer report on dose of treatment delivered using Fam-AID Fidelity Checklist. The checklist will measure extensiveness of treatment technique use on a 3-point scale from 0 = not at all to 2 = quite a bit/extensively. The checklist will be developed during the study pilot phase.
Family Involvement | Baseline to 6 months follow-up
  Family member session attendance in terms of number of sessions attended.
Internalizing disorder symptoms | Baseline to 6 months follow-up
  Adolescent and caregiver report on Revised Children's Anxiety and Depression Scale (RCADS). RCADS is a 47-item measure of youth's anxiety and depressive symptoms rated on a 4-point scale from 0 = Never to 3 = Always (range = 0 to 141). Higher numbers represent greater anxiety and depression.
Emotion Regulation | Baseline to 6 months follow-up
  Adolescent and caregiver report on Difficulties in Emotion Regulation Scale (DERS). DERS is a 16-item scale assessing difficulties with emotion regulation on a 5-point scale from 1 = almost never to 5 = almost always (range - . Higher numbers indicate greater difficulties regulating emotions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hogue A, Bobek M, Porter NP, MacLean A, Henderson CE, Jensen-Doss A, Diamond GM, Southam-Gerow MA, Ehrenreich-May J. Family Support Protocol for Adolescent Internalizing Disorders: Protocol for a Pre-Post Quantitative Treatment Development Study. JMIR Res Protoc. 2024 Sep 16;13:e64332. doi: 10.2196/64332. PMID 39284179